CLINICAL TRIAL: NCT06366204
Title: Determining Dietary Lysine Requirements in Healthy Lactating Women Using the Indicator Amino Acid Oxidation Technique
Brief Title: Lysine Requirements During Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H23-03119
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lactation; Breastfeeding, Exclusive; Breastfeeding
Keywords: Dietary Reference Intake; Lysine; Lactation; Indicator Amino Acid Oxidation; Lysine Requirements; Stable Isotopes
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Single day interventions; Repeated measures design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test Lysine Intake (Experimental): Randomly assigned one of 7 test lysine intakes that range from deficient to excess (12mg/kg/d to 84mg/kg/d). Participants may complete up to 4 study days, at different randomly assigned intakes.
  Interventions: Other: Dietary Lysine Intakes

INTERVENTIONS:
Other: Dietary Lysine Intakes — Participants consume 8 hourly meals that contain the assigned test lysine intake. Each meal will provide one-twelfth of the participants' daily energy requirements as estimated by 1.7 x Resting Energy Expenditure (REE) and adequate protein at 1.5 g.kg.d, to maintain a metabolic steady state. The meals are in the form of a crystalline amino acid protein shake, and nitrogenous free cookies.

SUMMARY:
The study aims to establish lysine requirements using the indicator amino acid oxidation (IAAO) method in women exclusively breastfeeding a single infant aged 3-4 months, and how maternal lysine needs change once infant transition to complimentary feeding at a later age of 9-10 months. Each 8-hour study day will have an assigned test lysine intake ranging from deficient to excess. The diets will be provided in a complete protein shake format, meeting all nutrient requirements except for the test lysine intake. Breath samples evaluate the indicator's oxidation to determine protein synthesis in response to lysine intake. Urine and one blood sample will be collected to assess metabolite concentrations.

DETAILED DESCRIPTION:
This study is a single-day intervention study where participants will be studied in a repeated measures design, with an individual having the option of participating in up 4 test lysine intakes for each lactation stage. A minimum of 10 women will be recruited, and the investigators hope to retain the same women for 8 study days to minimize data variability.

Potential participants will meet the researchers for a 1-hour preliminary assessment, where the investigators will evaluate their eligibility to participate in the study. During each study day, the participants will randomly receive a lysine test intake ranging from deficient to excess. The study day diets will consist of 8 hourly isocaloric and isonitrogenous meals in a protein shake, each presenting 1/12 of the daily energy requirement. The diets are composed of crystalline amino acid mixtures based on the composition of egg protein.

A Carbon-13 (13C) stable isotope tracer ( L-[1-13C]phenylalanine) will be added to the 5th-8th meal. The investigators will measure the rate of oxidation of this tracer expired in breath and the flux of this tracer by its enrichment in urine. The investigators will also collect a single blood sample to measure lysine metabolites. Lysine requirements will be determined by a two-phase linear regression crossover model on L-[1-13C]phenylalanine tracer oxidation using mixed-models regression to take repeated measures into account. The oxidation rate of the indicator amino acid exhibits a linear increase as the lysine intake rises until it reaches a plateau. The point at which this steady state is reached signifies that the test amino acid is predominantly utilized for protein synthesis. The primary endpoint is the lysine intake level at which the transition occurs from indicator oxidation (linear increase) to protein synthesis (plateau).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female
* 20-40 years
* Had a singleton pregnancy and is breastfeeding a single child.
* Exclusively breastfeeding an infant 3 - 4 months of age OR complimentary. feeding an infant 9-10 months of age.

Exclusion Criteria:

* Participants not in good health or have a history of metabolic, cardiovascular, neurological, genetic, endocrine, immune, or physical mobility disorders.
* Participants that had major pregnancy or delivery complications (e.g., preeclampsia/ eclampsia, placenta previa, postpartum haemorrhage, neonatal intensive care, gestational diabetes).
* Participants with substance dependence issues (e.g., nicotine, alcohol, marijuana, illicit drugs).
* Participants that have had breast surgery that may impact lactation, lactogenesis or breastfeeding.
* Participants that use medications that affect lactation (e.g. estrogenic birth control, anti-dopaminergic drugs, Methyldopa) or other continuous prescription medication.
* Participants with a pre-pregnancy BMI below 18 kg/m² or above 28 kg/m².
* Participants who are below 20 years of age or greater than 40 years of age.
* Infants' weight and length are under 3rd or above the 97th percentile, using the World Health Organization (WHO) percentile growth chart.
* Infants born before 38 weeks or after 42 weeks of gestation.
* Infants who use infant formula milk.
* Infants with known metabolic, cardiovascular, neurological, genetic, endocrine, immune, or physical mobility disorders.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Carbon 13 Oxidation | 8 hours
  Urine and breath samples will be collected to measure the rate of L-[1-13C]phenylalanine oxidation.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No